CLINICAL TRIAL: NCT05706428
Title: Cardiorespiratory Effects of Nasal High Frequency Ventilation in Moderate and Late Preterm Infants With Respiratory Distress
Brief Title: Cardiorespiratory Effects of Nasal High Frequency Ventilation in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Primary Investigator and Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0201417
Record Dates: First submitted 2023-01-21; First posted 2023-01-31 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Ventilator Lung; Newborn; Hemodynamic Instability; Echocardiography
Keywords: Premature infants; Echocardiography
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Nasal high-frequency ventilation (NHFV) group (case group):
  Interventions: Device: NHFOV
- Group II (Placebo Comparator): Nasal CPAP group (control group):
  Interventions: Device: NCPAP

INTERVENTIONS:
Device: NHFOV — The neonate patients with respiratory distress will have nasal high frequency ventilation as an initial mode of respiratory support.
  Arms: Group I
Device: NCPAP — The neonate patients with respiratory distress will have nasal continuous positive airway pressure as an initial mode of respiratory support.
  Arms: Group II

SUMMARY:
The aim of the present work is to study the cardio-respiratory effects of non-invasive ventilation (nasal high-frequency ventilation and nasal CPAP) as an initial therapy of respiratory distress in moderate and late preterm infants as regard:

I. Primary outcomes:

* Duration of the non- invasive respiratory support.
* Need of invasive ventilation in the first 72 hours.
* Short-term complications such as air leak syndromes, pulmonary hemorrhage, intraventricular hemorrhage, and nasal trauma.

II. Secondary outcomes:

* Need for surfactant administration.
* Days on invasive mechanical ventilation.
* Days on supplemental oxygen.
* Duration of hospital stay.
* Mortality rate. III. Hemodynamic changes during the period of non-invasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

Moderate and late preterm infants born between 32+0 to 36+6 weeks gestation(according to WHO definitions of preterm birth) admitted to the neonatal intensive care unit with spontaneous breathing and clinical manifestations of RD (tachypnea, nasal flaring, intercostal and subcostal retraction and or grunting).

Exclusion criteria:

* Any baby intubated for resuscitation or for other reasons.
* Obvious major congenital malformations or known complex congenital heart disease.
* Pulmonary hemorrhage.
* Cardiopulmonary arrest needing prolonged resuscitation.

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Superior vena cava blood flow in ml/kg/min | first 3 days of life
  The SVC diameter will be visualized from a high parasternal long axis view. The maximum and minimum internal diameters will be then measured. ✓ The SVC flow velocity will be visualized from a low subcostal view and the pulsed Doppler recording will be made at the junction of the SVC and the right atrium. ✓ SVC flow will be calculated using the method described by Kluckow and Evans:(27) SVC flow (ml/kg/min) = [VTI (cm/beat) × 3.14 × (mean SVC diameter2
  /4) × heart rate (beat/min)] Body weight in kg 11
Right ventricular output in ml /kg/min | first 3 days of life
  CSA (cm) (Cross sectional area of PV by long axis parasternal RV outflow view - 2D - immediately beneath pulmonary annulus
  - mid- systole - inner edge to inner edge) = π x (radius)2 ✓ VTI (cm) (Velocity Time Integral or Stroke Distance = Distance over which blood travels in once cardiac cycle → Long axis parasternal RV outflow view). ✓ SV (ml/beat) (Stroke Volume = CSA x VTI). ✓ Output (L/min.) COP = SV x HR.
left ventricular output in ml/kg/min | first 3 days of life
  CSA (cm) (Cross sectional area of AV by long axis parasternal view - 2D - immediately beneath aortic annulus - mid- systole - inner edge to inner edge) = π x (radius) 2 . ✓ VTI (cm) (Velocity Time Integral or Stroke Distance = Distance over which blood travels in once cardiac cycle → Apical 5- chamber view). ✓ SV (ml/beat) (Stroke Volume = CSA x VTI). ✓ Output (L/min.) COP = SV x HR
peak systolic velocity in anterior cerebral artery in cm/sec | first 3 days of life
  Trans-frontellar cranial sonography using Doppler study

CONTACTS AND LOCATIONS:
Overall Officials: Nader Abdelminem Fasseh, Study Director — Faculty of medicine, Alexandria University, Egypt; Mohamed Amen Hassan, MBChB, Principal Investigator — Faculty of medicine, Alexandria University, Egypt
Locations (1):
- Neonatal Intensive Care Unit (NICU) of Alexandria University Maternity Hospital., Alexandria, Egypt